CLINICAL TRIAL: NCT05154396
Title: Neratinib Dose Escalation Regimen for HER2 Positive Early Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese Academy of Medical Sciences (Other)
Responsible Party: Principal Investigator, Peng Yuan, Chief of VIP department, Chinese Academy of Medical Sciences
Organization: ChineseAMS (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NCC3075
Record Dates: First submitted 2021-10-09; First posted 2021-12-13 (Actual); Last update posted 2021-12-13 (Actual); Status verified 2021-11

CONDITIONS: HER2-positive Breast Cancer
MeSH Terms: interventions — neratinib

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Neratinib escalation 2 weeks（group A） (Experimental): Neratinib: 120mg/ day for days 1-7, 160mg/ day for days 8-14, and then 240mg/ day to complete 1-year treatment, or to tumor recurrence and metastasis, new breast cancer, or unacceptable adverse reactions within 1 year.
  Interventions: Drug: Neratinib
- Neratinib escalation 4 weeks（group B） (Experimental): Neratinib: 160mg/ day for days 1-14, 200mg/ day for days 15-28, and then 240mg/ day for 1 year, or to tumor recurrence and metastasis, new breast cancer, or unacceptable adverse reactions within 1 year.
  Interventions: Drug: Neratinib
- Neratinib standard dose control （group C） (Placebo Comparator): Neratinib: 240mg/ day for 1 year, or to tumor recurrence and metastasis, new breast cancer or unacceptable adverse reactions within 1 year.
  Loperamide prophylaxis: 4mg three times daily on days 1-14 and 4mg twice daily on days 15-56, followed by as needed, not exceeding 16mg/ day.
  Interventions: Drug: Neratinib

INTERVENTIONS:
Drug: Neratinib — Patients with her2-positive early breast cancer were treated with a dose escalation regimen of neratinib or a routine dose of neratinib combined with loperamide
  Other Names: Loperamide prophylaxis

SUMMARY:
This is a prospective study on the prevention of Neratinib-related diarrhea in a Chinese population, exploring the best options for reducing the incidence of neratinib-related diarrhea through either pharmacologic intervention (prophylactic antidiarrheal therapy) or non-pharmacologic intervention (dose escalation program).

DETAILED DESCRIPTION:
This is A prospective, randomized, single-center clinical trial, divided into 3 groups (experimental group: group A and group B, control group: group C), planned sixty patients were enrolled, with 20 patients in each group.

Experimental group: Group A (n=20) and group B (n=20) were given neratinib dose escalation regimen foranti-HER2 adjuvant therapy.In group A, the dose of neratinib climbed up to 240mg within 2 weeks, and in group B, the dose climbed up to 240mg within 4 weeks.

Control group: Group C (n=20) was given 240mg neratinib initially, but prophylactic loperamide antidiarrhea treatment was given at the same time within 2 months.

Diarrhea caused by neratinib often occurred within 1-2 months of initial treatment, so small dose of neratinib was used in both group A and group B at the time of initial treatment.

The incidence and severity of neratinib-related diarrhea in the three groups were observed, and DFS and other neratinib-related adverse events were followed up for a long time. The study is to evaluate the safety and efficacy of neratinib dose escalation regimen and conventional dose combined with loperamide regimen in enhanced anti-HER2 adjuvant therapy for early HER2-positive breast cancer.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 75 year-old women；
* ECOG score: 0-1；
* HER2 positive breast cancer diagnosed histologically is defined as HER2 (3+) by immunohistochemistry or HER2 (2+) with positive FISH test；
* Postoperative pathological stage ⅱ → ⅲ, or initial stage (before neoadjuvant therapy) ⅱ → ⅲ, radiographic assessment showed no metastasis;
* Complete 1 year of anti-HER2 therapy with trastuzumab, prior use of pertuzumab neoadjuvant + adjuvant therapy or T-DM1 adjuvant therapy is permitted;
* No major organ dysfunction, contraception;
* The patients have good compliance to the therapy and follow-up to be scheduled and are able to understand the study protocol and sign the Informed Consent Form.

Exclusion Criteria:

* Patients who are allergic to the study drug, cannot take the drug orally, or refuse the medication regimen;
* Prior treatment with TKI anti-HER-2 drugs (e.g. Lapatinib, Pyrotinib, etc.);
* Patients were enrolled in other studies or stopped taking other drugs within 4 weeks;
* Patients with serious dysfunction of important organs (heart, liver and kidney);
* Patients with other malignancies, other than cured non-melanoma skin cancer, carcinoma in situ of the cervix and other tumors that have been cured for at least 5 years;
* In pregnancy, lactation patients;
* In the active stage of other acute or chronic infectious diseases;
* The patients have uncontrollable mental illness;
* There is a known history of human immunodeficiency virus;
* There are other circumstances in which the investigator suggested that the patient should not participate in the study.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Primary Endpoint | up to 3 year after the last patient enrolled
  Incidence of grade ≥3 diarrhea in patients with her2-positive early breast cancer treated with neratinib dose escalation versus neratinib conventional dose combined with loperamide

SECONDARY OUTCOMES:
Secondary Endpoint | up to 3 year after the last patient enrolled
  3-year invasive disease-free survival (iDFS%) and other safety events

CONTACTS AND LOCATIONS:
Overall Officials: Peng Yuan, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences